CLINICAL TRIAL: NCT04909684
Title: Dose Tapering and Early Discontinuation to InCreAse cosT-effectIveness Of Immunotherapy for Non-small Cell Lung Carcinoma
Brief Title: Dose Tapering and Early Discontinuation to InCreAse cosT-effectIveness Of Immunotherapy for NSCLC
Acronym: DEDICATION-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Society of Physicians for Pulmonology and Tuberculosis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVALT30 / DEDICATION-1; 2020-000493-15 (EudraCT Number)
Record Dates: First submitted 2021-04-26; First posted 2021-06-02 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-07

CONDITIONS: NSCLC
Keywords: pembrolizumab; immunotherapy; biomarkers; dose tapering
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): 100% pembrolizumab
- Intervention (Experimental): 75% pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — The approved doses of 400 mg every 6 weeks (Q6W) and 200 mg every 3 weeks (Q3W) will be decreased to a 300 mg Q6W dose. The approved dose of 150 mg Q3W will be decreased to a 100 mg Q3W dose.
  Arms: Intervention

SUMMARY:
Rationale: Immune checkpoint inhibitors have shown to improve the overall survival for patients with metastasized non-small cell lung carcinoma (NSCLC) but the optimal dosing and patient selection are still a matter of discussion. The pembrolizumab dose, for instance, may be reduced significantly without decreasing treatment efficacy. Furthermore, as approximately only half of all patients responds to treatment, there is an urgent need to develop (early) treatment response prediction markers to select those who benefit from treatment.

Objective: Primary: to investigate the non-inferiority of pembrolizumab 75% versus pembrolizumab 100% in terms of overall survival. Secondary: to develop biomarkers that predict immunotherapy treatment response.

Study design: An open label randomized non-inferiority study.

Study population: 750 patients with NSCLC, eligible for treatment with pembrolizumab, in line with the current ESMO clinical practice guidelines.

Intervention: Patients will be randomized to standard of care (100%) versus reduced dose (approx. 75%, depending on treatment schedule) pembrolizumab.

Main study parameters/endpoints: One-year overall survival rate

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

1.1 General introduction The recent introduction of immune checkpoint inhibitors (ICI) has dramatically changed treatment and prognosis of metastasized non-small cell lung carcinoma (NSCLC). Depending on the type of treatment, the line of treatment and tumour characteristics, response rates of 20 to over 60% are shown, and durable responses are seen. However, the accessibility to novel cancer treatments in The Netherlands is at serious risk due to the rising incidence of cancer as well as the exponentially increasing costs of these new and effective drugs. As an example, the yearly costs for treatment of metastasized NSCLC with Pembrolizumab single agent therapy in the Netherlands was estimated to be 27 million euro in 2018. With the recent new indications in the first line treatment in lung cancer alone this sum is surpassed by at least a four-fold. With ever increasing strains on healthcare budgets, we have a societal responsibility to decrease treatment costs wherever possible. Furthermore, for the individual patient it is very relevant to offer a treatment only if it is effective. By investing in a more tailored treatment we intend to personalize treatment, thereby allowing significant cost-reduction, without reducing the promise that all these new treatment options hold for the individual patients. For the individual patient we have the responsibility to expose patients to no more drug than strictly necessary and to limit the number of hospital visits.

1.2 Immune checkpoint inhibitors ICI have revolutionized systemic treatment of many malignancies. By targeting the programmed death (ligand)-1 (PD-1/PD-L-1) axis with specific ICI's, T-cell tolerance can be overcome and cellular immune response to tumour cells is boosted. In contrast to previous treatment modalities, ICI are able to induce durable responses thereby improving overall survival in NSCLC. In 2015, nivolumab was the first PD1 monoclonal antibody that showed a clinically relevant efficacy in patients with metastasized disease. Since then, many phase III trials have shown positive results thereby improving both progression free and overall survival in patients with advanced and or metastasized disease. ICI's have been introduced rapidly in The Netherlands and the efficacy results of real-life data are comparable to those from phase 3 trials. Both PD1 and PDL1 monoclonal antibodies are currently approved for the treatment of NSCLC and, at present, the vast majority of patients fit for systemic treatment will receive a form of ICI.Currently, pembrolizumab forms the mainstay first line therapy for metastasized NSCLC. We expect that in the Netherlands approximately 2500-3000 NSCLC patients will be treated with an immune checkpoint inhibitor on a yearly basis, with pembrolizumab as the cornerstone in treatment.

1.3 Dose tapering of immune checkpoint inhibitors There are no known exposure-toxicity relationships for pembrolizumab and usually dosing regimens are usually developed for prescriber's convenience, i.e. as a one-dose-fits-all regimen. During clinical phase development a dose is selected that will result in therapeutic exposure in all patients, indicating that in the majority of patients pembrolizumab is overdosed.

1.4 Pembrolizumab dose tapering rationale As pembrolizumab will be the main ICI for NSCLC in the upcoming years, we focus on pembrolizumab in the current study. We postulate that the approved dose of pembrolizumab (200 mg every three weeks [Q3W] or 400 mg every 6 weeks [Q6W]) can be decreased to a 300 mg dose Q6W or 100 mg dose Q3W without compromising efficacy.

1.4.1 Dose development and pharmacokinetic-pharmacodynamic relationships of pembrolizumab in NSCLC

An initial phase I trial of pembrolizumab demonstrated complete peripheral PD-1 target engagement at a dose of 1 mg/kg, which was continued for more than 21 days. Furthermore, no difference in pharmacodynamics were observed at doses of 1, 3, or 10 mg/kg. Also, linear pharmacokinetics were observed from doses of 0.3 mg/kg and up. This indicated saturation of target-mediated clearance and, thus, complete peripheral PD-1 blockade at doses of 0.3 mg/kg and higher. Lastly, no dose-limiting toxicities were observed at the 0.3 to 10 mg/kg dose levels and no apparent relationship between dose and toxicity was observed at these dose levels. Mechanism-based translational models of intratumor exposure of this study further suggested robust clinical activity at doses of 2 mg/kg Q3W. The preclinical dose development was supported by clinical pharmacokinetic/pharmacodynamic modelling of the ex-vivo IL-2 stimulation ratio response. If the PD-1 blockade is complete, this ratio decreases to a minimum of 1. It was shown that from doses of 1 mg/kg Q3W and higher, and serum concentrations of 1 ug/ml and higher, the pharmacodynamic response (measured as target engagement or IL-2 stimulation ratio) reached a plateau (1). From the dose finding studies, it was decided that the 2 mg/kg Q3W dose was carried forward for further clinical development. Although the 2 mg/kg Q3W dosing regimen was eventually authorized by the FDA to treat advanced NSCLC following first-line therapy, recently a fixed 200 mg Q3W dose was introduced and used in more recent trials, like the KEYNOTE-024 study. More recently, Merck has proposed to administer a 400 mg Q6W dosing regimen, based on population pharmacokinetic and pharmacodynamic simulations and the Committee for Medicinal Products for Human Use (CHMP) of the European Medicines Agency (EMA) has recommended the approval of this dosing regimen on March 4th 2019. The change of drug label for the 200 mg Q3W and the 400 mg Q6W dosing regimens was based on in-silico investigations only, using previously developed population pharmacokinetic and pharmacodynamic models of pembrolizumab in cancer patients. It was predicted that a weight-based 2 mg/kg dosing regimen did not relevantly reduce pharmacokinetic variability and that the pharmacokinetic exposure of a 200 mg Q3W dose or 400 mg Q6W flat dose resulted in similar or higher exposure than the approved 2 mg/kg dose for all indications. Notably, it was shown that a flat dose of approximately 150 mg Q3W resulted in bioequivalent exposure as the clinically proven effective and safe dose of 2 mg/kg. Although the 200 mg Q3W and 400 mg Q6W dosing regimens resulted in a higher exposure than associated with the clinically proven effective and safe dosing regimen of 2 mg/kg Q6W, the exposure was lower than found for the 10 mg/kg Q2W dose, which was just as safe as the 2 mg/kg Q3W dose. The 200 mg Q3W and 400 mg Q6W regimens were, therefore, considered equivalent to the previously approved 2 mg/kg Q3W dosing regimen in terms of efficacy and safety. In short, the above data indicate that pembrolizumab at its current dose (200 mg Q3W or 400 mg Q6W) is overdosed and can be tapered safely, because:

1. Linear pharmacokinetics of pembrolizumab are observed at doses of 0.3 mg/kg Q3W and higher. Linear pharmacokinetics indicate that receptor-mediated clearance of the therapeutic antibody does not take place due to saturation of the receptor at the concentrations associated with the 0.3 mg/kg dose.
2. A plateau in pharmacodynamic response is observed at doses of 1 mg/kg and higher, which translates to that a flat dose of approximately 75 mg Q3W or 150 mg Q6W is as effective as the currently approved dosing regimens of 200 mg Q3W and 400 mg Q6W.
3. The lowest proven clinically effective dose of pembrolizumab for treatment of NSCLC is 2 mg/kg and the currently approved dosing regimens of 200 mg Q3W or 400 mg Q6W result in higher exposure than associated with the 2 mg/kg Q3W regimen, indicating that the dose can be safely reduced.

2. OBJECTIVES

Primary Objective:

- To investigate the non-inferiority of reduced dose pembrolizumab versus standard of care for treatment of advanced stage NSCLC in terms of overall survival.

Secondary Objective(s):

* To develop immune checkpoint inhibitor response biomarkers.
* To study possible effect modification from co-medication on treatment outcome.

  3. STUDY DESIGN The current study will be an open label non-inferiority trial of reduced dose pembrolizumab versus standard of care (administered with or without chemotherapy), either as monotherapy or in combination with chemotherapy in NSCLC patients who are eligible for treatment with a pembrolizumab-based regimen.

3.1 Dedication-1 can be classified as a low intervention clinical trial

Many clinical trials pose only a minimal additional risk to subject safety compared to normal clinical practice. According to the EU clinical trial regulation 536/2014, these low-intervention clinical trials are of crucial importance for assessing standard treatments and diagnoses, thereby optimizing the use of medicinal products and thus contributing to a high level of public health. Trials like these should be subject to less stringent rules, like monitoring, requirements for the contents of the master file and traceability of investigational medicinal products. The published scientific evidence supporting the safety and efficacy of an investigational medicinal product not used in accordance with the terms of the marketing authorization could include high quality data published in scientific journal articles, as well as national, regional or institutional treatment protocols, health technology assessment reports or other appropriate evidence.We consider the current study a low intervention clinical trial in line with the definition from the EU clinical trial regulation 536/2014 for the following reasons:

* In the proposed study, the investigational medicinal product is authorized. Also, the use and dose of pembrolizumab are supported by solid evidence from the EMA approval data of pembrolizumab with the same level of evidence that was used for registration of the 200 mg Q3W and the 400 mg Q6W dosing regimens. Furthermore, the lower dose is already used routinely in some institutions in the Netherlands.
* The additional diagnostic and monitoring procedures besides the treatment with the investigational product do not pose more than minimal risk. This is fully in line with EU clinical trial regulation 536/2014 definition of a low intervention clinical trial.
* Low intervention clinical trials as defined in the regulation according to the "expert group on clinical trials for the implementation of Regulation (EU) No 536/2014" should fall within categories A and B as defined by the OECD. We conclude that our study falls in category B "Modified use" and is, therefore, a low interventional clinical trial. The OECD framework supports the risk-adapted approach by introducing a stratified approach that is based on the marketing authorization status of the medicinal product being investigated, with a trial-specific approach.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care.
* Participants must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
* Subjects with cytologically or histologically confirmed advanced stage or recurrent NSCLC (per the 8th International Association for the Study of Lung Cancer classification, eligible for treatment of NSCLC with pembrolizumab in line with ESMO guidelines.
* Prior adjuvant or neoadjuvant chemotherapy is permitted as long as the last administration of the prior regimen occurred at least 3 months prior to enrolment.
* Prior chemoradiation for locally advanced disease is also permitted as long as the last administration of chemotherapy or radiotherapy (which ever was given last) occurred at least 3 months prior to enrolment.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Males and Females, ages 18 years (or age of majority) and older.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
* Women must not be breastfeeding.
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of 5 months (30 days of ovulatory cycle plus the time required for the investigational drug to undergo five half-lives).
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of 7 months (90 days plus the time required for pembrolizumab to undergo five half-lives) after the last dose of investigational drug. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Subjects with symptomatic untreated CNS metastases are excluded. Subjects are eligible if CNS metastases are asymptomatic and / or adequately treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrolment.In addition, participants must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to treatment assignment.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications (see list below) within 14 days of enrolment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted.
* a CD4+ T-cell count of less than 100 cells/μL
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* History of allergy or hypersensitivity to study drug components.
* Subjects may not have previously received a solid organ transplantation.
* Total body weight <40 or >140 kg
* Absence of or unknown PD-L1 status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
One-year overall survival rate | At least one year or until death, whichever comes first.
  Percentage of patients alive after one year.

SECONDARY OUTCOMES:
Median overall survival | At least one year or until death, whichever comes first.
  The length of time from the start of treatment that half of the patients are still alive.
Two-year overall survival rate | At least one year or until death, whichever comes first.
  Percentage of patients alive after two years.
Best overall response rate | At least one year or until death, whichever comes first.
  Best overall response at the end of treatment will be summarized by treatment arm for all eligible, treated subjects. The summary table will include counts and percentages for each response category (CR, PR, SD, PD, unevaluable) as reported by the investigator
Disease control rate | At 3, 6 and 12 months
  Percentage of patients who have achieved complete response, partial response and stable disease after 3, 6 and 12 months.
Duration of treatment | At least one year or until death, whichever comes first.
  From start of treatment (pembrolizumab/chemotherapy) until end of treatment (as reported in CRF).
EQ-5D questionnaire | at baseline, 3, 6 and 12 months
  Quality of life, measured with the validated EuroQol Five Dimensions Health Questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Michel vd Heuvel, prof., Principal Investigator — Head of Department
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands